CLINICAL TRIAL: NCT03459040
Title: A Proof of Concept Pilot Trial of Alpha-1-Antitrypsin for Pre-Emption Of Steroid-Refractory Acute GVHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: John Levine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, John Levine, Professor of Internal Medicine and Pediatrics, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GCO 17-2666; P01CA039542 (NIH)
Record Dates: First submitted 2018-03-02; First posted 2018-03-08 (Actual); Results first posted 2021-05-24 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Graft-versus-host-disease; GVHD
MeSH Terms: conditions — Graft vs Host Disease | interventions — alpha 1-Antitrypsin

STUDY DESIGN:
Intervention Model Description: Open label single arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- alpha-1-antitrypsin (AAT) (Experimental): 16 doses of AAT through a catheter placed into a blood vessel over eight weeks.
  Interventions: Drug: Alpha 1-Antitrypsin

INTERVENTIONS:
Drug: Alpha 1-Antitrypsin — AAT will be given either in the hospital or the outpatient clinic two times per week.
  Other Names: AAT

SUMMARY:
Bone marrow transplant (BMT) patients can develop graft-versus-host disease (GVHD), a serious and potentially fatal complication. The researchers have developed a blood test to identify patients most at risk for developing severe GVHD. Patients who consent to this study will have their blood tested up to two times after BMT to determine if they are at high risk for severe GVHD. The tests will be performed one week and two weeks after BMT. Patients who are high risk will be treated with a drug called alpha-1-antitrypsin (AAT) to see if it prevents the development of severe GVHD. Patients will receive 16 doses of AAT through a catheter placed into a blood vessel over eight weeks. AAT will be given either in the hospital or the outpatient clinic two times per week. Patients will be followed for the development of severe GVHD for up to four months from the BMT and will continue to be followed at routine clinic visits for up to one year after BMT.

ELIGIBILITY:
Inclusion Criteria:

* High risk prediction score as determined by the Mount Sinai Acute GVHD International Consortium (MAGIC) algorithm at either day 7 or day 14 post Hematopoietic cell transplant (HCT).
* Any donor type (e.g., related, unrelated) or stem cell source (bone marrow, peripheral blood, cord blood).
* Donor and recipient match each other for at least 7/8 HLA-loci (HLA-A, B, C, and DR)
* Any conditioning regimen (non-myeloablative, myeloablative, or reduced intensity) is acceptable.
* GVHD prophylaxis must include a calcineurin inhibitor combined with methotrexate or mycophenolate.
* The use of serotherapy to prevent GVHD (e.g., antithymocyte globulin) prior to day 3 post-HCT is permitted
* Direct bilirubin must be <2 mg/dL unless the elevation is known to be due to Gilbert syndrome within 3 days prior to enrollment.
* ALT/SGPT and AST/SGOT must be <5 x the upper limit of the normal range within 3 days prior to enrollment.
* Signed and dated written informed consent obtained from patient or legal representative.

Exclusion Criteria:

* Patients who develop acute GVHD prior to start of study drug
* Patients at very high risk for relapse post HCT as defined by very high disease risk index
* Patients participating in a clinical trial where prevention of GVHD is the primary endpoint
* Uncontrolled active infection (i.e., progressive symptoms related to infection despite treatment or persistently positive microbiological cultures despite treatment or any other evidence of severe sepsis)
* Patients who are pregnant
* Patients on dialysis within 7 days of enrollment
* Patients requiring ventilator support or oxygen supplementation exceeding 40% FiO2 within 14 days of enrollment.
* Patients receiving investigational agent within 30 days of enrollment. However, the Principal Investigator (PI) may approve prior use of an investigational agent if the agent is not expected to interfere with the safety or the efficacy of alpha-1-antitrypsin.
* History of allergic reaction to alpha-1-antitrypsin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2020-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Levine, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (5):
- United States (5):
  - City of Hope, Duarte, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Ohio State University, Columbus, Ohio
  - Vanderbilt University, Nashville, Tennessee

REFERENCES:
- [Result] Gergoudis SC, DeFilipp Z, Ozbek U, Sandhu KS, Etra AM, Choe HK, Kitko CL, Ayuk F, Aziz M, Baez J, Ben-David K, Bunworasate U, Gandhi I, Hexner EO, Hogan WJ, Holler E, Kasikis S, Kowalyk SM, Lin JY, Merli P, Morales G, Nakamura R, Reshef R, Rosler W, Srinagesh H, Young R, Chen YB, Ferrara JLM, Levine JE. Biomarker-guided preemption of steroid-refractory graft-versus-host disease with alpha-1-antitrypsin. Blood Adv. 2020 Dec 22;4(24):6098-6105. doi: 10.1182/bloodadvances.2020003336. PMID 33351103

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited and enrolled between August 2018 and July 2019.
Groups:
- Alpha-1-antitrypsin (AAT): AAT was administered intravenously at a loading dose of 90 mg/kg (study day 0), followed by twice weekly doses of 45 mg/kg for 15 more doses (totaling 16 doses over 8 weeks).
Period: Overall Study
Arm/Group | Alpha-1-antitrypsin (AAT)
Started | 30
Completed | 21
Not Completed | 9
Not completed — Death | 8
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Alpha-1-antitrypsin (AAT)
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 51 [20 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Diagnosis [Count of Participants; unit: Participants]
  Myelodysplastic syndrome | 13
  Acute myelogenous leukemia | 9
  Acute lymphoblastic leukemia | 5
  Nonmalignant disease | 2
  Non-Hodgkin's lymphoma | 1
Donor [Count of Participants; unit: Participants]
  Matched related | 3
  Matched unrelated | 26
  Mismatched related | 0
  Mismatched unrelated | 1
GVHD Prophylaxis [Count of Participants; unit: Participants] — Chronic Graft Vs. Host Disease
  Participants
    CNI/MTX - calcineurin inhibitor/methotrexate | 14
    CNI/MMF -Calcineurin inhibitors/mycophenolate mofetil | 0
    calcineurin inhibitor/sirolimus | 15
    Cyclophosphamide based | 0
    Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of High Risk Patients Who Develop Steroid Refractory GVHD
Description: Number of High Risk patients who develop steroid refractory GVHD by day 100 post Hematopoietic cell transplant (HCT) .
  Steroid refractory GVHD defined as patients who did not achieve Complete Response (CR) or Partial Response (PR) by day 28 of systemic steroid treatment OR if additional immunosuppression beyond steroids was given for treatment of GVHD prior to 28 days of steroid treatment.
  * CR: All evaluable organs (skin, liver, GI tract) stage 0. For a response to be scored as CR on day 28, the patient must be in CR on that day and have had no intervening additional GVHD therapy.
  * PR: An improvement in one or more organ involved with GVHD symptoms without worsening in others. For a response to be scored as PR on day 28, the patient must be in PR on that day and have had no intervening additional GVHD therapy.
Time Frame: Day 100 post HCT.
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha-1-antitrypsin (AAT)
Number analyzed (Participants) | 30
Participants | 6

2. Secondary Outcome: Number of Participants Alive at 6 Months and 1 Year
Description: Overall survival - The number of that patients are still alive from the start of treatment at 6 months and 1 year
Time Frame: 6 months and 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha-1-antitrypsin (AAT)
Number analyzed (Participants) | 30
Participants
  6 months | 26
  1 year | 22

3. Secondary Outcome: Number of Participants With Non-relapse Mortality (NRM)
Description: Number of participants with NRM - deaths which could not be attributed to disease relapse or progression. Non-relapse mortality defined as death without prior relapse.
Time Frame: 6 months and 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha-1-antitrypsin (AAT)
Number analyzed (Participants) | 30
Participants
  6 months | 3
  1 year | 6

4. Secondary Outcome: Number of Participants With Relapse
Description: Number of participants with relapse at one year. Relapse defined as recurrence of disease that required transplant.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha-1-antitrypsin (AAT)
Number analyzed (Participants) | 30
Participants | 3

5. Secondary Outcome: Number of Participants With Clinically Relevant GVHD States Grade II-IV GVHD
Description: Number of participants with clinically relevant GVHD states grade II-IV GVHD requiring systemic treatment.
  GVHD grades II-IV are defined as
  * Rash covering more than 50% of the body surface area, AND/OR
  * Total bilirubin > 2 mg/dl AND/OR
  * Persistent nausea or vomiting, AND/OR
  * Diarrhea > 500 ml/day AND/OR
  * Severe abdominal pain requiring treatment or blood present in the diarrhea
Time Frame: 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha-1-antitrypsin (AAT)
Number analyzed (Participants) | 30
Participants | 12

6. Secondary Outcome: Number of Participants Achieving Overall Response
Description: For patients who develop GVHD prior to day 100 post-HCT, the number of participants achieving overall response. The overall response rate = complete remission and partial remission (CR + PR) 28 days after initiation of systemic steroid treatment.
Time Frame: Day 28
Population: This is the number of patients who developed GVHD and were systemically treated (not all patients on study developed GVHD and of those that did develop GVHD, not all received systemic treatment).
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha-1-antitrypsin (AAT)
Number analyzed (Participants) | 16
Participants | 10

7. Secondary Outcome: Number of Participants With Severe GI GVHD Stage 3 or 4
Description: Number of participants with severe GI GVHD stage 3 or 4. GI GVHD stage 3 or 4 is defined as diarrhea >1000 ml/day OR severe abdominal pain requiring treatment OR blood present in the diarrhea.
Time Frame: By day 100 post-HCT
Measure: Count of Participants; unit: Participants
Groups:
- Number of Participants Requiring Steroid Treatment: Number of participants with chronic GVHD requiring systemic steroid treatment
  alpha-1-antitrypsin (AAT) AAT was administered intravenously at a loading dose of 90 mg/kg (study day 0), followed by twice weekly doses of 45 mg/kg for 15 more doses (totaling 16 doses over 8 weeks).
Arm/Group | Number of Participants Requiring Steroid Treatment
Number analyzed (Participants) | 30
Participants | 4

8. Secondary Outcome: Number of Participants With Chronic GVHD Requiring Systemic Steroid Treatment
Description: Number of participants with chronic GVHD requiring systemic steroid treatment. Chronic GVHD Requiring Systemic Steroid Treatment: defined as the development of symptoms of chronic GVHD according to NIH Consensus Criteria that require treatment with oral or intravenous corticosteroids.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha-1-antitrypsin (AAT)
Number analyzed (Participants) | 30
Participants | 8

9. Secondary Outcome: Number of Participants With Serious Infections
Description: Number of participants with serious infections (defined as grade 3 by the Blood and Marrow Transplant Clinical Trials Network). Serious Infection: Defined as bacterial, fungal, viral or parasitic infections that required oral or intravenous treatments such as antibiotics.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha-1-antitrypsin (AAT)
Number analyzed (Participants) | 30
Participants | 2

ADVERSE EVENTS:
Time Frame: up to 1 year
Arm/Group | Alpha-1-antitrypsin (AAT)
All-Cause Mortality (participants affected / at risk) | 8/30
Serious Adverse Events (participants affected / at risk) | 14/30
Other Adverse Events (participants affected / at risk) | 9/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alpha-1-antitrypsin (AAT) (N=30)
Engraftment Syndrome (General disorders) | 1
GVHD (Immune system disorders) | 4 — Graft Versus Host Disease
Headache (Nervous system disorders) | 1
Line Infection: Gram negative Bacilli-Citrobacter (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1 (1)
Fungal Infection: Pneumocystis carinii pneumonia (PCP) (Infections and infestations) | 1 — Pneumocystis carinii pneumonia
Fungal Infection: Aspergillus (Infections and infestations) | 1
Bronchopulmonary hemorrhage (DAH) (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 2
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Relapse (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alpha-1-antitrypsin (AAT) (N=30)
Atrial Fibrillation (Cardiac disorders) | 1
Maculopapular rash with engraftment syndrome (Skin and subcutaneous tissue disorders) | 1
Oral mucositis (Gastrointestinal disorders) | 1
Maculopapular Rash (Skin and subcutaneous tissue disorders) | 1
Hypertension (Cardiac disorders) | 1
Klebsiella (Infections and infestations) | 1
Infusion Reaction (Injury, poisoning and procedural complications) | 5
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Generalized muscle weakness (General disorders) | 1
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Hyponatremia (Blood and lymphatic system disorders) | 1
Hyperglycemia (Blood and lymphatic system disorders) | 1
Low platelets (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/40/NCT03459040/Prot_SAP_000.pdf